CLINICAL TRIAL: NCT05214599
Title: A Phase I/II, Multicenter, Double-blind, Parallel, Randomized Trial to Assess Pharmacokinetics, Efficacy, Tolerability and Safety of Different Budesonide Oral Gel Doses in Adults Subjects of Both Genders With Eosinophilic Esophagitis (EoE)
Brief Title: Pharmacokinetics, Efficacy, Tolerability and Safety of Different Budesonide Oral Gel Doses in Adults' Subjects of Both Genders With Eosinophilic Esophagitis (EoE)
Acronym: BESIDE
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Business decision
Sponsor: Bazell Pharma AG (Industry)
Responsible Party: Sponsor
Organization: Amzell (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BAZ006-001
Record Dates: First submitted 2022-01-03; First posted 2022-01-28 (Actual); Last update posted 2024-08-23 (Actual); Status verified 2024-08

CONDITIONS: Eosinophilic Esophagitis
MeSH Terms: conditions — Eosinophilic Esophagitis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group 1 (Experimental): Low dose
  Interventions: Drug: Budesonide Gel
- Group 2 (Experimental): Middle dose
  Interventions: Drug: Budesonide Gel
- Group 3 (Experimental): High dose
  Interventions: Drug: Budesonide Gel

INTERVENTIONS:
Drug: Budesonide Gel — Twice daily regimen

SUMMARY:
A phase I/II, multicenter, double-blind, parallel, randomized trial to assess pharmacokinetics, efficacy, tolerability and safety of different budesonide oral gel doses in adults subjects of both genders with eosinophilic esophagitis (EoE)

ELIGIBILITY:
Inclusion Criteria:

* Subjects able to read, understand and sign the Informed Consent Form (ICF) approved by Ethical Committee;
* Male and female subjects aged between 18 and 75 years old;
* Body weight between 60-100 kg;
* Body mass index (BMI) ≥ 18.5 and ≤ 29.9 kg/m2;
* Non-childbearing potential female subjects. Childbearing potential is defined as: post-menopausal women (defined as 12 months of amenorrhea or more), hysterectomized women, oophorectomized (bilateral) women and/or those who underwent tubal ligation;
* Female participants of childbearing potential who test negative for the pregnancy test on the day of administration of the first dose of the drug (Visit 1), as well as throughout the clinical trial;
* Female participants who practice adequate contraception or who abstain from all activities that could result in pregnancy for at least 28 days before administering the first dose of the drug (Visit 1);
* Female participants who agree to continue adequate contraception for 1 month after administration of the last dose of the investigational drug;
* Participants diagnosed with EoE, verified from a combination of symptoms compatible with EoE and histological finding greater than 15 eosinophils per high-power field in at least one esophageal mucosal biopsy;
* Participants unresponsive to stable dose of proton-pump inhibitor (PPI).

Exclusion Criteria:

* Subjects with a malignancy history within the last 5 years, except from successfully treated basal cell carcinoma;
* History of esophageal stenosis requiring dilation and/or stenosis at endoscopy not allowing to pass the endoscope;
* Subjects with a eosinophilic gastroenteritis diagnosis (presence of eosinophilic infiltrate in gastric antrum and duodenum);
* Subjects with a reflux esophagitis history;
* Subject with a previous serious asthma diagnosis;
* Subjects with a gastroesophageal tract disease that, at the investigator's discretion, is deemed as an obstacle to take part in the trial;
* People with chronic diseases on regular drugs that, in the investigator's opinion, may interfere with the trial;
* Medical conditions such as serious heart or lung diseases preventing the safe performance of endoscopy;
* Subjects with conditions known to be related to esophageal eosinophilia, including Crohn's disease, Churg-Strauss, achalasia and hypereosinophilic syndrome;
* Subjects who have been on oral, intranasal or systemic corticosteroid at least 15 days prior to trial start;
* Smoker of having quit smoking less than 6 months ago;
* Have a history of excessive alcohol intake for at least 6 months prior to trial start (intake of 5 or more alcoholic beverages in one day or 15 or more alcoholic beverages per week);
* Subjects having 5 or more cups of tea or coffee per day and who cannot abstain from them for the trial period;
* Be on CYP3A4 inhibitors, such as ketoconazole and grapefruit juice;
* Electrocardiogram (ECG) findings that, in the investigator's opinion, may jeopardize participation in the trial;
* History or presence of gastrointestinal or liver disease or other condition interfering with drug absorption, distribution, excretion or metabolism;
* Subjects with hypersensitivity or contraindication of using any formulation components;
* Subjects who have been part of trial protocols in the last 12 (twelve) months (CNS Resolution 251, dated August 7, 1997, item III, sub-item J);
* Have donated blood (> 500 mL) or undergone major surgery within the 3 months prior to the ICF signature date;
* Have been vaccinated for the 30 days prior to admission;
* Clinical evidence of infectious process potentially contributing for dysphagia (candidiasis, cytomegalovirus (CMV), herpes);
* Other dysphagia cause identified at endoscopy (peptic stenosis, web, ring, achalasia, esophageal neoplasm);
* Breastfeeding subjects, who plan to become pregnant or with a positive pregnancy test during the trial;
* Any medical condition or laboratory change that, in the investigator's opinion, may jeopardize participation in the trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-04-23 (Actual); Primary Completion 2024-11 (Estimated); Study Completion 2025-04 (Estimated)

PRIMARY OUTCOMES:
Determination of Pharmacokinetic Profiles | First 24 hours after a single drug dose administration
  Peak Plasma Concentration (Cmax)
Determination of Pharmacokinetic Profiles | First 24 hours after a single drug dose administration
  Area under the plasma concentration versus time curve (AUC)
Determination of Pharmacokinetic Profiles | First 24 hours after a single drug dose administration
  Half-life (T1/2)
Determination of Pharmacokinetic Profiles | First 24 hours after a single drug dose administration
  Oral clearance (CL/F)
Proportion of subjects reaching a histological response | 8 weeks of treatment
  ≤ 6 eosinophils per high power field
Improvement in dysphagia symptoms consistent with the disease | 8 weeks of treatment
  EAT (Eating Assessment Tool) -10 questionnaire

SECONDARY OUTCOMES:
Assessment of non-serious and serious adverse events rate | Through 8 weeks
Quality of life assessment of subjects | Through 8 weeks
  WHOQOL-bref questionnaire

IPD SHARING:
Plan to Share IPD: No
There is not a plan to make individual participant data (IPD) available